CLINICAL TRIAL: NCT03269877
Title: Hypersplenism in Patients With Liver Cirrhosis and Portal Hypertension: Prevalence, Pattern, Correlations, and Therapy
Brief Title: Hypersplenism in Patients With Liver Cirrhosis and Portal Hypertension
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ramy Mahmoud Fathy Elbarody, Principal investigator at Tropical Medicine and Gastroenterology Department, Assiut University
Other Study IDs: HSLC
Record Dates: First submitted 2017-08-28; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Hypersplenism
MeSH Terms: conditions — Hypersplenism

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver cirrhosis and hypersplenism: Patients proven to have Liver Cirrhosis and Hypersplenism based on clinical examination, Laboratory findings, and abdominal ultrasound examinaton

SUMMARY:
The spleen could be considered a neglected organ. To date, it has been deemed an ancillary organ in portal hypertension or an organ localization in lymphoproliferative diseases. Hypersplenism is a common disorder characterized by an enlarged spleen which causes rapid and premature destruction of blood cells. It can result from any splenomegaly. It is most common with splenomegaly secondary to portal hypertension and hematological disorders. Portal Hypertension is an important cause of splenomegaly in most tropical countries This work will involve a series of studies aiming to:

1. Assess the prevalence and pattern of hypersplenism, and grade the severity of cytopenias in patients with cirrhosis and portal hypertension.
2. Elucidate the relationship between hypersplenism, in these patients, and:

   1. The severity of liver cirrhosis as assessed by Child's and the Model of End-stage Liver Disease (MELD) scores.
   2. The presence and grade of gastroesophageal varices as assessed by upper endoscopy.
   3. The presence of hepatocellular carcinoma
   4. Portal hemodynamics and portal vein thrombosis as assessed by Doppler Ultrasound.
3. Test the hypothesis that leucopenia in cirrhotic patients may be caused, at least in part, by apoptosis of polymorphnuclear leucocytes.

DETAILED DESCRIPTION:
Hypersplenism is a clinical syndrome characterized by: (1) Splenomegaly (2) Pancytopenia or a reduction in the number of one or more types of blood cells (3) Normal production or hyperplasia of the precursor cells in the marrow or a so called maturation arrest (4) Decreased red blood cells survival (5) Decreased platelet survival. In hypersplenism, its normal function accelerates, and begins automatically to remove cells that may still be normal in function. It can be classified into three categories: I) Primary hypersplenism; II) Secondary hypersplenism; III) Occult hypersplenism. A number of mechanisms causing hypersplenism have been identified, and mainly involve retention in the spleen, phagocytosis, and autoimmunity.

PMN have a short life-span and spontaneously undergo apoptosis in the living body. Although neutropenia in cirrhotic patients is associated with the presence of splenomegaly and increased clearance of granulocytes in the spleen, the complete sequence of events leading to neutropenia in cirrhosis is at present unknown. Although neutrophils are programmed to undergo apoptosis at the time of differentiation, the rate of apoptosis is under the regulation of external factors. Therefore, changes in the rate of PMN apoptosis are likely to occur in the setting of cirrhosis. The rate of apoptosis and its contribution in in cirrhotic patients with or without neutropenia and hypersplenism need further evaluation.

Hypersplenism is a common complication in patients with chronic liver diseases, leading to decreases in platelet and hemoglobin levels, and correlates with the severity of cirrhosis. Splenomegaly is often used radiologically as an indicator of cirrhosis. Moreover, one study has shown that hypersplenism is more frequent and more severe in younger cirrhotic patients, and another one has addressed that platelet count to spleen diameter ratio non-invasively identifies severe fibrosis and cirrhosis in patients with chronic hepatitis and cirrhosis. Many studies also investigated the relationship between size of gastroesophageal varices and platelet count/spleen diameter ratio in cirrhotic patients which was found that it could be used as also a non-invasive indicator of esophageal varices. Indeed, there is little published on the actual frequency of hypersplenism.

Hypersplenism is correlated with increased risk of hepatocellular carcinoma in post-hepatitis cirrhosis. One study addressed that several factors including hypersplenism in post hepatitis cirrhosis may contribute to hepatocellular carcinoma development. It also addressed the efficiency of splenectomy in reducing hepatocellular carcinoma risk. Another study concluded that microwave ablation of the spleen combined with partial hepatectomy is a safe and effective technique for treatment of hepatocellular carcinoma and hypersplenism.

It has been shown that portal venous pressure positively correlates with spleen size. Duplex-Doppler has been employed in pathophysiological investigations of portal hemodynamics and is accepted as the first-line imaging technique in patients with suspected portal circulation disorders, particularly in portal hypertension. The measurement of the hepatic venous pressure gradient has served as the gold standard for assessing the degree of portal hypertension, however, due to its invasive nature and the requirements for skilled expertise and special equipment, some Ultrasound indices, such as Hepatic Vein and Portal Vein indices, exhibited an increased accuracy for diagnosing portal hypertension. These indices may be useful in clinical practice for the detection of significant portal hypertension.

To date, no studies have fully assessed these correlations of hypersplenism in the same cirrhotic patients, which can be useful in diagnostic aspects, assessment, grading of severity, therapeutic interventions or even leading to the development of a new scoring system for hypersplenism.

ELIGIBILITY:
Inclusion Criteria:

* All patients with documented evidence of liver cirrhosis (of any etiology other than alcoholic cirrhosis) and portal hypertension, based on clinical examination, abdominal ultrasound examination, upper gastrointestinal endoscopy.
* Male and female patients aged between 18-60 years.

Exclusion Criteria:

* Patients with splenomegaly of any cause other than liver cirrhosis.
* Patients with any lymphoproliferative disorders.
* Patients with extrahepatic malignancy.
* Patients younger than 18 years old.
* Any associated cardiovascular disease.
* Failure to obtain consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All admitted patients who fulfill the inclusion criteria over a period of one year will be included. We are expecting that a total of 400 patients will be recruited.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence | 6 months
  Percentage of hypersplenism in patients proven to have liver cirrhosis and portal hypertension
Severity | 1 year
  Depending mainly on the severity of cytopenia of the blood elements (RBCs, WBCs, and platlets), hypersplenism will be graded as mild, moderate, or severe, and given a total score of <2 points, 2-3 points, and >3 points, respectively

SECONDARY OUTCOMES:
Correlations with severity of liver disease | 1 year
  Percentage of hypersplenism patients, falling into each category of the Child-Pugh score for assessment of severity of liver disease (A, B, or C)
Correlation with Eosophageal varices | 1 year
  Percentage of hypersplenism patients in each category of grades of oesophageal varices (small, moderate, or large)
Correlations with hepatocellular carcinoma | 1 year
  Percentage of hypersplenism patients having hepatocellular carcinoma

REFERENCES:
- [Result] Kim G, Cho YZ, Baik SK, Kim MY, Hong WK, Kwon SO. The accuracy of ultrasonography for the evaluation of portal hypertension in patients with cirrhosis: a systematic review. Korean J Radiol. 2015 Mar-Apr;16(2):314-24. doi: 10.3348/kjr.2015.16.2.314. Epub 2015 Feb 27. PMID 25741193
- [Result] Lv Y, Lau WY, Li Y, Deng J, Han X, Gong X, Liu N, Wu H. Hypersplenism: History and current status. Exp Ther Med. 2016 Oct;12(4):2377-2382. doi: 10.3892/etm.2016.3683. Epub 2016 Sep 7. PMID 27703501
- [Result] McCormick PA, Walker S, Benepal R. Hypersplenism is related to age of onset of liver disease. Ir J Med Sci. 2007 Dec;176(4):293-6. doi: 10.1007/s11845-007-0089-8. Epub 2007 Oct 18. PMID 17943410
- [Result] Orlando R, Lirussi F, Basso SM, Lumachi F. Splenomegaly as risk factor of liver cirrhosis. A retrospective cohort study of 2,525 patients who underwent laparoscopy. In Vivo. 2011 Nov-Dec;25(6):1009-12. PMID 22021698
- [Result] Ramirez MJ, Titos E, Claria J, Navasa M, Fernandez J, Rodes J. Increased apoptosis dependent on caspase-3 activity in polymorphonuclear leukocytes from patients with cirrhosis and ascites. J Hepatol. 2004 Jul;41(1):44-8. doi: 10.1016/j.jhep.2004.03.011. PMID 15246206